CLINICAL TRIAL: NCT05723276
Title: Probing the Functional Magnetic Resonance Imaging Response to Psilocybin in Functional Neurological Disorder (PsiFUND)
Brief Title: Psilocybin in Functional Neurological Disorder
Acronym: PsiFUND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TBC
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2024-10

CONDITIONS: Functional Neurological Disorder
MeSH Terms: conditions — Conversion Disorder | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Experimental): Psilocybin with therapeutic support
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Psilocybin 25mg PO

SUMMARY:
The goal of this study is to learn about the brain network response in people who have functional neurological disorder who are administered with a single dose of the psychedelic psilocybin with therapeutic support.

The main question it aims to answer is:

Can the default mode network, a brain network thought to be relevent in FND, be modified by the administration of psilocybin based on functional magnetic resonance imaging before and after the dose?

ELIGIBILITY:
Inclusion Criteria:

1. Age 25 - 60 years.
2. Fluent in the English language
3. A diagnosis of FND from a neurologist and/or neuropsychiatrist as per DSM-5 criteria
4. Moderate or severe symptoms (≥4 on Clinical Global Impression Severity (CGI-S) scale) which have been present for >12 months and have failed to respond to best available treatment.
5. Able to tolerate fMRI scanning procedures.

Failed to respond is defined as an inadequate response to a full course of FND-specific therapy, including psychological therapy (cognitive behavioural therapy) or physiotherapy. Either therapy must have been undertaken by a suitably trained expert in FND and must have been specifically targeted at FND symptoms.

Exclusion Criteria:

1. Diagnosis of severe depression (defined as meeting DSM-5 criteria) on the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
2. Diagnosis of bipolar affective disorder (defined as meeting DSM-5 criteria for bipolar I or bipolar II) on the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
3. Diagnosis of a psychotic disorder (defined as meeting DSM-5 criteria) on the MINI 7.0, EXCEPT substance/medication induced psychotic disorder where the duration was limited to the acute period of direct intoxication with the substance/medication. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
4. Diagnosis of drug or alcohol dependence disorder (defined as meeting DSM-5 criteria) on the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
5. Diagnosis of a personality disorder (defined as meeting DSM-5 criteria) on the MINI 7.0. Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
6. Diagnosis of any dementia (defined as meeting DSM-5 criteria for any dementia disorder) based on clinical interview by a psychiatrist.
7. Diagnosis of any autistic spectrum disorder (defined as meeting DSM-5 criteria for any dementia disorder) based on clinical interview by a psychiatrist.
8. Diagnosis of any learning disability (defined as meeting DSM-5 criteria for any dementia disorder) based on clinical interview by a psychiatrist
9. Significant suicidal behaviour in past 12-months defined using the Columbia-Suicide Severity Rating Scale (C-SSRS) and confirmation based on clinical interview by a psychiatrist
10. Any other factor which would render the participant unsuitable for psilocybin and/or interfere with a supportive therapeutic relationship and/or preclude safe follow-up.
11. Those unable to give informed consent
12. Medical diagnosis incompatible with psilocybin treatment (see Section 8.2.1)
13. Inability to provide a screening blood sample, urine sample or electrocardiogram.
14. Biochemical abnormalities (defined as falling outside the normal reference range) as evaluated by a full blood count, full biochemistry profile and thyroid function tests. Biochemical abnormalities must also be determined as clinically significant by a medical doctor to fulfil the criterion for exclusion.
15. Electrocardiographic abnormalities, defined as any abnormality that is not normal sinus rhythm and determined as clinically significant by a medical doctor.
16. Women of childbearing potential not using contraception.
17. Pregnant or breast-feeding women.
18. Non-registration with a GP or failure to consent to sharing of the GP summary care record and any psychiatric assessments held.
19. Those enrolled in another clinical or research study.
20. Use of any psychedelic substances >2 times in past 12 months.
21. Any factor which would exclude the participant from magnetic resonance imaging (e.g., presence of metal)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in functional connectivity in default mode network | One week prior dosing versus one week post dosing (intra-subject)

CONTACTS AND LOCATIONS:
Locations (1):
- South London and Maudsley NHS Foundation Trust, London, United Kingdom